CLINICAL TRIAL: NCT03249012
Title: Comparing the Quality of Life Associated With Empiric Calcium Repletion and Parathormone (PTH) Based Calcium Repletion for Post Thyroidectomy Hypoparathyroidism
Brief Title: Quality of Life Related to Different Treatment Protocols for Post-thyroidectomy Hypoparathyroidism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Jean-Philippe Vézina, Otolaryngologist and Head & Neck Surgeon, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-3422
Record Dates: First submitted 2017-08-09; First posted 2017-08-15 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Hypoparathyroidism Postprocedural; Quality of Life
MeSH Terms: interventions — Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empiric calcium and calcitriol repletion group (Experimental): All patients in this group will receive post-operative calcium carbonate and calcitriol.
  Interventions: Other: Empiric use of Calcium Carbonate and Calcitriol
- PTH based repletion group (Experimental): Patients in this group will be prescribed calcium carbonate and calcitriol based on their post-operative PTH.
  Interventions: Other: PTH based Calcium Carbonate and Calcitriol repletion

INTERVENTIONS:
Other: Empiric use of Calcium Carbonate and Calcitriol — Empiric calcium carbonate and calcitriol repletion
  Arms: Empiric calcium and calcitriol repletion group
Other: PTH based Calcium Carbonate and Calcitriol repletion — PTH based treatment
  Arms: PTH based repletion group

SUMMARY:
This study aims to compare two different protocols commonly used in the management of post thyroidectomy hypoparathyroidism : PTH based calcium repletion and empiric repletion. The investigators aim to compare the quality of life associated with these two protocols in a randomized trial.

DETAILED DESCRIPTION:
Enrolled patients will be randomized in two treatment groups. In group 1, all patients will receive calcium carbonate and calcitriol in the post-operative period, with standardized weaning. In group 2, patients will be prescribed calcium carbonate and calcitriol only if their post-operative PTH dosage is 25% or less of the pre-operative dosage, or if post-operative PTH is inferior to 15.

The Short-Form 36 (SF-36) questionnaire (French canadian version) will be used to assess quality of life pre-operatively and at post-op week 1 and 4. Symptoms of hypocalcemia and adverse effects of calcium carbonate and calcitriol will be monitored at week 1 and 4.

ELIGIBILITY:
Inclusion Criteria:

* Total thyroidectomy or completion hemithyroidectomy

Exclusion Criteria:

* Need for neck dissection
* Unable to fill in questionnaires (intellectual deficit, severe psychiatric disorder, illiterate, does not speak French or English)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline quality of life at 1 and 4 weeks | Pre-op, 1 week post-op and 4 weeks post-op
  Short Form 36 (SF-36) questionnaire

SECONDARY OUTCOMES:
Occurence and change in pharmacologic adverse effects of calcium carbonate and calcitriol | 1 week post-op, 4 weeks post-op
  A questionnaire about the adverse effects of calcium carbonate and calcitriol will be completed at post-op week 1 and 4
Occurence and change in symptoms of hypocalcemia | 1 week post-op, 4 weeks post-op
  A questionnaire about symptoms of hypocalcemia will be completed at post-op week 1 and 4.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Quebec, Québec, Quebec, Canada